CLINICAL TRIAL: NCT07375732
Title: Transcranial Electrical Stimulation for Noninvasive Study of Menopausal/Perimenopausal Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Pulkit Grover, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: STUDY2025_00000313
Record Dates: First submitted 2026-01-20; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Menopausal Depression; Menopause Hot Flashes; Menopause; Menopause Related Conditions
Keywords: Noninvasive Neuromodulation; Transcranial Electrical Stimulation; Depression; Vasomotor Symptoms; Hot Flashes
MeSH Terms: conditions — Depression; Hot Flashes | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation of Occipital Cortex (Sham Comparator): Transcranial Electrical Stimulation will be delivered to the occipital cortex (mapped using the 10 20 EEG system) at a similar current/pain level as the active stimulation trial.
  Interventions: Device: Transcranial Electrical Stimulation
- Motor Cortex Stimulation (Experimental): Transcranial electrical stimulation will be delivered to the primary motor cortex (mapped using the 10-20 EEG system) and current will be injected such that there are evoked motor potentials in the distal extremities.
  Interventions: Device: Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Transcranial Electrical Stimulation — SharpFocus transcranial electrical stimulation (TES) uses a multichannel stimulator connected to a scalp electrode to deliver precisely timed, intensity-modulated electrical pulses. By varying the timing, amplitude, and location of these pulses, the system achieves focal stimulation of targeted cortical regions.
  Investigators will use Digitimer DS8R and/or Digitimer DS5 current stimulators to apply all current stimuli. These stimulators are CE certified and are intended for use in human research applications. The stimulator safely delivers brief duration (50-2000µs) current pulses for transcranial electrical stimulation and activation of nerves and muscles via surface electrodes. The current output of the DS8R is adjustable over the range 0mA to 1000mA, with a compliance voltage of up to 400V and an energy limit of 300mJ.

SUMMARY:
Participants are being invited to a research study. This research aims to assess the tolerability of transcranial electrical stimulation of the brain, and explore the response of TES on menopausal/perimenopausal symptoms including hot flashes effects, depression/anxiety, memory-problems, and muscular problems. This study will assess what types of electrical brain stimulation affect different menopausal related symptoms. This study will help guide the development of electrical stimulation to be used for improving women's health during menopause transition.

DETAILED DESCRIPTION:
The purpose of this study is to assess the tolerability of transcranial electrical stimulation of the brain, and explore the response of TES on menopausal/perimenopausal symptoms including vasomotor effects , depression/anxiety, memory-problems. Electrical stimulation comprises a pattern of electrical currents that are delivered into the skin non-invasively using an array of electrodes adhered to the skin surface. Pain administration and sensory testing may be performed using thermodes, which are devices attached to limbs whose temperature is controlled using a computer (heat and cold pain). Temperature will be varied across time and heat/cold delivered to assess any changes in self-reported pain and/or non-invasive Electroencephalography (EEG) and functional Near-Infrared Spectroscopy (fNIRS). Examining the association of locations of current delivery with changes in self-reported pain and EEG/fNIRS recordings will help assess the spatiotemporal dynamics in the brain relevant to pain perception and the nature of their effects on pain (e.g. increase or decrease). Prior to testing the effects on pain, the individual's primary motor cortex may be localized by delivering short pulses at locations close to the motor cortex and measuring muscle responses using electromyography (EMG) electrodes placed on muscles (e.g. on the arms and legs).

The participant's resting state and pain-evoked brain activity will also be recorded using non-invasive Electroencephalography (EEG) and functional Near-Infrared Spectroscopy (fNIRS).

The stimulation techniques - called SharpFocus Transcranial Electrical Stimulation (SharpFocus TES) - consist of patch arrays (a set of electrodes arranged in a grid and embedded in a flexible substrate that conforms to the skin surface) or individual electrodes being installed at various locations including the head, arms, and legs. Some of the electrodes on the scalp inject current for brain stimulation. The rest of the electrodes are for recording. Conductive cream, gel, or hydrogel is placed between the electrode and skin to improve adhesion and conductivity. Additionally, or alternatively, classic cup (e.g. gold-cup) electrodes (10 mm diameter or 6 mm diameter), used routinely in the clinic, might also be used, especially for participants with thick or long hair. A multichannel electrical stimulator connects to the electrode array to deliver pulses of electrical current that are varied in timing, intensity, and location to allow fine-grained control of the site(s) of stimulation in the brain.

For sensory effects, participants will be asked to report any modulation of pain sensation they feel on electrical stimulation. Experiments will be performed to measure effects on muscle activity and perceived sensations.

Results from these experiments will be used to verify and refine computational models that have been developed to simulate biophysical effects of SharpFocus TES. Furthermore, it will aid in the understanding of how the central nervous system affects several of the symptoms seen in menopause/perimenopause. The ultimate goal of this research is to create a wearable interface that can stimulate parts of the cortex for a variety of applications pertaining to menopause/perimenopause.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 60 years
* Participants falling under stages -2 to +2 in the Stages of Reproductive Aging Workshop (STRAW +10) as defined below:
* Early menopause transition (Stage -2): Increased variability in menstrual cycle defined as persistent difference of 7 days or more in the length of consecutive cycles. Persistence is defined as recurrence within 10 cycles of the first variable cycle.
* Late menopause transition (Stage -1): Occurrence of amenorrhea of 60 days or longer.
* Final Menstrual Period (Stage 0): Have undergone 12 consecutive months without a menstrual period, not due to other medical causes.
* Early Postmenopause (Stage +1): 5-8 years after final menstrual period.
* Late Postmenopause (Stage +2): >8 years after final menstrual period.
* Participants having frequent hot flashes (at least once a day).

Exclusion Criteria:

* Disorders that may mask or coincide with menopause and peri-menopause, such as: Primary Ovarian Insufficiency, Thyroid disease (Hyper/hypothyroidism), Hyperprolactinemia, Cushing's syndrome, Endometrial/Ovarian Cancer, Polycystic Ovary Syndrome (PCOS), Functional hypothalamic amenorrhea
* Concurrent drugs:
* GnRH agonist/antagonist
* Tamoxifen/aromatase inhibitors
* Other conditions: Recent hematoma (<48 hours), History of hemorrhagic disorders (any platelet disorder (ITP, TTP, HUS, Glanzmann thrombasthenia), Hemophilia A/B, history of arterial insufficiency, any prior history of malignancy, current pregnancy, a lifetime history of severe, uncontrolled mood disorders (anxiety, depression, bipolar), psychotic disorders, other neural disorders, or heart disease, any condition that makes them unable to perform tasks outlined in experiment, tattoos on sensory testing sites.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Depression | From enrollment to the end of treatment at 22 days
  Menopause related depression will be queried using the Menopause Depression Rating Scale (Meno-D) questionnaire as well as the CES-D inventory prior to and at the end of each arm. The Meno-D is a 12-item self-report or clinician-rated scale specifically developed to assess depression during the perimenopausal transition. It captures unique symptom clusters such as irritability, memory issues, low energy, and somatic complaints not typically addressed in general depression scales. The minimum score is 0 and the maximum is 48 points.Between 20-24 points is considered to denote mild perimenopausal depression, needing onward monitoring. Between 24-32 points suggests moderate perimenopausal depression needing treatment. At 32 points and above, the woman is considered to have severe perimenopausal depression needing treatment.
Sleep Quality | Study enrollment to end of study at 22 days
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a widely used self-report questionnaire that assesses overall sleep quality and disturbances over the past month. It includes 19 items grouped into seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Total global score ranges from 0 to 21. Higher scores indicate poorer sleep, with a total score above 5 suggesting significant sleep impairment.
Menopause Quality of Life | Upon enrollment to 22 days
  Quality of life will be measured using the Menopause rating scale (MRS) survey. The MRS is a validated, self-administered tool designed to assess health-related quality of life in midlife women. It measures the severity of 11 common menopausal symptoms across three domains: psychological, somato-vegetative, and urogenital to evaluate symptom burden and changes over time, including before and after treatment. Scores range from 0 to 44 with 0 being no menopausal symptoms and 44 being severe menopausal symptoms.
Center for Epidemiological Studies-Depression Inventory (CES-D) | Upon enrollment to 22 days
  General depressive symptoms will be measured with the Center for Epidemiological Studies-Depression Inventory (CES-D). The CES-D is a 20-item self-report measure designed to assess depressive symptoms experienced over the past week. Items cover mood, somatic complaints, and interpersonal difficulties, with responses rated on a 4-point scale. Higher total scores reflect more severe depressive symptoms, with a score of 16 or above suggesting risk for clinical depression. The scale ranges from a minimum of 0 (indicating very low depression) to a maximum of 60 (indicating high depressive symptoms).
Numerical Rating Scale | Upon enrollment to 22 days
  A numerical rating scale (NRS) uses numbers to quantify subjective experiences of pain. NRS scores will be self-reported on a scale of 0-10 with 0 being no pain and 10 being worst pain imaginable. NRS will be presented to patients during calibration phases of Transcranial Electrical Stimulation (TES), during heat pain thresholding, and during pressure pain thresholding in the form of a visual scale and be asked to vocalize a number between 0 and 10 in response to a pain stimulus.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | Upon enrollment to 22 days
  Measures of catastrophic thinking related to pain will be measured with the Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report questionnaire widely used self-report tool that measures catastrophic thinking related to pain. It assesses three domains-rumination, magnification, and helplessness based on thoughts and feelings about pain, even when not currently in pain. Total scores range from 0-52, where higher scores indicate greater catastrophizing; a total score above 30 indicates a clinically significant level.
Impulsive Behavior Scale | Upon enrollment to 22 days
  Measures of impulsivity will be measured with the UPPS Inventory. The UPPS is a 59-item self-report questionnaire developed to assess four distinct facets of impulsivity: urgency, lack of premeditation, lack of perseverance, and sensation-seeking. Grounded in the Five Factor Model of personality, it integrates items from multiple established impulsivity scales. Responses are rated on a 4-point Likert scale, with higher scores indicating greater impulsive tendencies. Higher scores indicate greater impulsivity, with subscale minimums/maximums ranging from 4 to 16.
Brief Pain Inventory | Upon enrollment to 22 days.
  Daily pain severity will be measured with the Brief Pain Inventory (BPI). The BPI is a self-report questionnaire assessing pain severity and its interference with daily functioning. Respondents rate pain intensity (worst, least, average, current) and interference with activities (e.g., mood, work, sleep) on 0-10 scales. Scores yield severity and interference indices, with higher values indicating greater pain impact. The BPI demonstrates strong reliability, validity, and sensitivity across diverse clinical populations.
Electromyography Recording | Upon enrollment to 22 days
  High density electromyography (HD-EMG) will be recorded in response to transcranial electrical stimulation (TES) throughout the study period. HD-EMG and/or bipolar EMG electrodes will be placed on the participant's limbs or torso muscles to record resulting activity. EMG activity is recorded in microvolts and resulting motor evoked potentials (MEPs) will be quantified in terms of changes in amplitude (root mean square ratio), shape, and latency.
Sternal Skin Conductance | Upon enrollment to 22 days
  A galvanic skin response (GSR) will be recorded at the sternum during in person experiments throughout the experimental and sham periods for detection of hot flashes. GSR will be recorded with a TMSi GSR sensor attached to disposable Ag/Cl electrodes. Measurements will be recorded in microsiemens and the presence of hot flashes during the experimental session will be characterized in terms of amplitude, duration, and frequency.
Functional Near-Infrared Spectroscopy | Upon enrollment to 22 days
  Functional near-infrared spectroscopy (fNIRS) will be recorded to measure blood flow changes during the study period. Data collection will use the NIRSport 2 system (NIRx Medical Technologies), a portable, wearable fNIRS device. A custom optode array embedded in an elastic, swimmer's-cap-style headpiece will be positioned to record from bilateral frontal and parietal cortices, including the prefrontal cortex and primary somatosensory cortex. The optode array consists of emitter and detector optodes connected to the NIRSport 2 system via flexible fiberoptic cables. Emitter optodes deliver low-intensity near-infrared light at 690 nm and 830 nm. Adjacent detector optodes collect the fraction of light not absorbed by cortical tissue and return it to the instrument for conversion to optical density. From these signals, concentrations of oxygenated hemoglobin (HbO, 830 nm) and deoxygenated hemoglobin (HbR, 690 nm) are estimated using the modified Beer-Lambert law.
Electroencephalogram | Upon enrollment to 22 days
  Electroencephalogram (EEG) signals will be measured throughout the study period prior to the start of stimulation. To record EEG an investigator will use an EEG instrument made by BioSemi Corporation (ActiveTwo EEG system) and/or a BrainVision system. An elastic cap supports an array of up to 32 gold-cup EEG electrodes (1cm diameter). Each electrode contains a metal tip connected to a small amplifier inside a plastic box. After being amplified with a dense array of amplifiers, EEG signals from each electrode are digitized by an integrated digital EEG computer system. Measured in micovolts, this EEG signal will be characterized to look for any changes in oscillatory power bands (alpha, beta, theta, delta) using spectral density analsyis.
Heat Pain Thresholding | Upon enrollment to 22 days
  A thermode system placed on the distal forearm will be used to determine sensitivity to heat pain throughout the study period. Medoc and QST Lab thermode systems will be used for administering pain using heat and cold. Hot or cold temperatures (0-50 °C) will be applied for short periods of time (<60 sec). Then, to individualize the noxious temperature used to elicit offset analgesia, a heat/cold pain calibration procedure is performed to determine the temperature that produces 50/100 pain on the computerized numerical rating scale. For calibration, a series ascending heat/cold steps that are each ~30 seconds long with a break (interstimulus interval, ISI) between steps of ~2 minutes. Responses to pain are recorded. After reaching a temperature that elicits a 50/100, the heat/cold pain calibration procedure is stopped and this temperature is referred to as T1. The site of testing on the body will include the forearm, thumb, and trapezius depending on the specific
Pressure Pain Thresholding | Upon enrollment to 22 days
  A digital pressure algometer will be used to apply mechanical pressure to the base of the thumb throughout the study period. The experimenter will manually apply the pressure at a rate of 1lbf/s. From this the pressure pain threshold will be calculated and defined as the minimum amount of force that induces pain by the subject

IPD SHARING:
Plan to Share IPD: Yes